CLINICAL TRIAL: NCT05697198
Title: PRospective REgistry of Advanced Stage CancER (PREFER) Patients to Assess Prevalence of Actionable Biomarkers and Driver Mutations Using the OmniSeq Test and Creation of a Biobank from Community Cancer Clinics in the United States to Address Disparities in Precision Medicine
Brief Title: PRospective REgistry of Advanced Stage CancER (PREFER) Patients to Assess Prevalence of Actionable Biomarkers and Driver Mutations to Address Disparities in Precision Medicine
Acronym: PREFER
Status: Completed | Type: Observational
Sponsor: Labcorp Corporation of America Holdings, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: PREFER
Record Dates: First submitted 2022-12-21; First posted 2023-01-25 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer; Ovarian Cancer; Uterine Cancer; Colorectal Cancer; Stomach Cancer; Esophageal Cancer; Pancreatic Cancer; Melanoma; Breast Cancer; Head and Neck Cancer; Soft Tissue Sarcoma; Rhabdomyosarcoma; Prostate Cancer
MeSH Terms: conditions — Lung Neoplasms; Ovarian Neoplasms; Uterine Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Pancreatic Neoplasms; Melanoma; Breast Neoplasms; Head and Neck Neoplasms; Sarcoma; Rhabdomyosarcoma; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — In the optional biobank component of the study, participants may elect to give a blood sample that will be stored in cell-free DNA streck tubes for future research use
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (8):
- Cohort lung cancer
  Interventions: Diagnostic Test: OmniSeq Test
- Gyn malignancies
  Interventions: Diagnostic Test: OmniSeq Test
- Gastrointestinal malignancies Cohort
  Interventions: Diagnostic Test: OmniSeq Test
- Melanoma Cohort
  Interventions: Diagnostic Test: OmniSeq Test
- Breast cancer Cohort
  Interventions: Diagnostic Test: OmniSeq Test
- Head and neck cancer Cohort
  Interventions: Diagnostic Test: OmniSeq Test
- Sarcoma and soft tissue cancer cohort
  Interventions: Diagnostic Test: OmniSeq Test
- Prostate cancer
  Interventions: Diagnostic Test: OmniSeq Test

INTERVENTIONS:
Diagnostic Test: OmniSeq Test — Genomic and immune profiling assay for all solid tumors

SUMMARY:
The objective of this Study is to collect, process, and transfer biologic samples such as blood and/or tissue biopsies to determine the concordance of detected alterations obtained through liquid biopsy analyses compared to next generation sequencing of time-matched or archival tissue specimens from individuals with advanced solid tumors.

Examples of locally advanced and metastatic tumors include stage III and IV cancers (ex. lung, breast, all gastrointestinal malignancies, all gynecologic malignancies, prostate cancer, head and neck tumors, soft tissue cancers, and melanoma). These specimens will be analyzed for diagnostic purposes and research (either by Labcorp/OmniSeq or to a third-party recipient designated by Labcorp/OmniSeq). Labcorp/OmniSeq may transfer the specimens and data to its clients, including commercial, academic or non-profit research institutions; or alternatively, may retain the specimens in its repository for future research use at the sole discretion of Labcorp/OmniSeq and or assignees. Labcorp/OmniSeq will maintain all detailed clinical information including demographic data (de-identified), ethnicity, disease state, stage (radiological, pathological and clinical-whichever is relevant).

DETAILED DESCRIPTION:
The scope of this pilot includes increasing uptake of personalized medicine (PM) testing using the OmniSeq test for identifying actionable target mutations in clinically appropriate patients and improving the quality of care particularly in practices providing care to minority and underserved patient populations. The research scope of this pilot covers 3 major areas that are necessary to understand the feasibility and best approaches.

i. How to identify appropriate steps and strategies to improve compliance to achieve optimum testing for all cancer patients, including all minority patients, in accordance with approved guidelines.

ii. How to contact, trace and test all eligible patients and impact outcomes to prevent future cancers in unaffected relatives

iii. Impact of trace back approach to identify, test, and guide appropriate clinical management and intervention in patients already diagnosed with eligible cancer types who have not yet been tested. This can be done by: 1) searching pathology records or tumor registry databases 2) community engagement campaigns and 3) self-referral based on family (and/or personal) cancer history.

The PREFER Registry will enable Labcorp/OmniSeq to create a biorepository in addition to a registry. The benefits are as follows:

* The biorepository registry will collect clinical data, store biological specimens, and maintain additional associated information for future use in research.
* The biorepository will address healthcare disparities by increasing representative samples of tissues available for research from community oncology practices to reflect ethnicity and social determinants of health (SDOH). The biorepository would create catalogs of different mutations and/or germline information in different ethnicities for future drug development.
* The biorepository will ensure the quality of data, enhance research, and manage the accessibility and distribution/disposition of biospecimens in its collection.
* The biorepository will develop a tissue bank for serious malignant disorders with appropriate clinical data points that will support the development of newer molecules for targeted therapy. This will facilitate expansion of indications of existing molecules by providing better understanding of RNA/DNA derived anomalies and diseases as well as response criteria.

Contribution to Science:

* The PREFER registry and biorepository would collect clinical data, maintain biological specimens, and associated information, for future use in research.
* The biorepository would address healthcare disparities representing samples of biospecimens for the research from rural population

The seven steps to establish and operationalize of Labcorp/Omniseq biorepository:

1. Informed consent (includes permission to commercialize use of specimens at a future date to develop drugs at the sole discretion of Labcorp/OmniSeq)
2. Data Collection: All relevant clinical information will be entered in a central data repository. Data will include a unique identifier, demographic data, as well as all data points discussed previously
3. Sample collection: Since patient will be undergoing standard diagnostic work up for suspected primary malignant disorder as a standard course of action at the point of care (POC) facility, the registry will not be adding any additional invasive clinical or diagnostic intervention
4. Sample Processing/Shipping and Handling (Per SOP)
5. Electronic Case Report From (ECRF) and data point to be entered by POC Facility
6. Storage or inventory
7. Retrieval, Redistribution of biological specimens

ELIGIBILITY:
Case Inclusion Criteria

* Any gender, race, or ethnicity is acceptable
* Must be at least 18 years of age
* All subjects must fall into the following group:

All Cases will be classified as following cohorts

Cohort lung cancer - Subject must meet the following criteria:

* Recently diagnosed advanced lung cancer
* Locally advanced and metastatic solid tumors
* Treatment naïve (not yet treated or tumor removed; biopsy acceptable) and/or on treatment
* Previously Treated: If treated, must have developed resistance and testing will be looking at change in therapy based on results of testing

Gyn malignancies (list ovarian and uterine cancer separately)

* Recently diagnosed advanced gynecological malignancies
* Locally advanced and metastatic solid tumors
* Treatment naïve (not yet treated or tumor removed; biopsy acceptable).
* Previously Treated: If treated, must have developed resistance and testing will be looking at change in therapy based on results of testing

Gastrointestinal malignancies Cohort (list all cancers separately-colorectal, gastric, esophageal and pancreatic)

* Recently diagnosed advanced gastrointestinal malignancy
* Locally advanced and metastatic solid tumors
* Treatment naïve (not yet treated or tumor removed; biopsy acceptable).
* Previously Treated: If treated, must have developed resistance and testing will be looking at change in therapy based on results of testing

Melanoma Cohort

* Recently diagnosed advanced melanoma
* Locally advanced and metastatic solid tumors
* Treatment naïve (not yet treated or tumor removed; biopsy acceptable).
* Previously Treated: If treated, must have developed resistance and testing will be looking at change in therapy based on results of testing

Breast cancer Cohort

* Recently diagnosed advanced breast cancer
* Locally advanced and metastatic solid tumors
* Treatment naïve (not yet treated or tumor removed; biopsy acceptable).
* Previously Treated: If treated, must have developed resistance and testing will be looking at change in therapy based on results of testing

Head and neck cancer Cohort

* Recently diagnosed advanced head and neck cancer
* Locally advanced and metastatic solid tumors
* Treatment naïve (not yet treated or tumor removed; biopsy acceptable).
* Previously Treated: If treated, must have developed resistance and testing will be looking at change in therapy based on results of testing

Sarcoma and soft tissue cancer cohort

* Recently diagnosed advanced cancer
* Locally advanced and metastatic solid tumors
* Treatment naïve (not yet treated or tumor removed; biopsy acceptable).
* Previously Treated: If treated, must have developed resistance and testing will be looking at change in therapy based on results of testing

Prostate cancer

* Recently diagnosed advanced cancer
* Locally advanced and metastatic solid tumors
* Treatment naïve (not yet treated or tumor removed; biopsy acceptable).
* Previously Treated: If treated, must have developed resistance and testing will be looking at change in therapy based on results of testing

Additional Requirements

* Subjects must be diagnosed by appropriate histopathology
* Subjects can have any concurrent diseases
* Must voluntarily sign and understand the most current Institutional Review Board/Independent Ethics Committee (IRB/IEC) - approved Informed Consent Form (ICF) prior to study participation. Witness must sign the informed consent form if the subject is illiterate.

Exclusion Criteria

* Subjects incapable of understanding the items listed in the ICF and the consent process
* Pregnant females
* Subjects with a history of or known psychiatric illness that deems them unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with advanced solid tumors
Sampling Method: Probability Sample
Enrollment: 1429 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The percent adoption of the OmniSeq next generation sequencing (NGS) testing platform in an advanced cancer patient population compared to baseline over a 2 year period | 2 years

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Clinical Site, Fort Payne, Alabama
  - Clinical Site, Orange City, Florida
  - Clinical Site, Stuart, Florida
  - Clinical Site, Dublin, Georgia
  - Clinical Site, Fort Wayne, Indiana
  - Clinical Site, Covington, Louisiana
  - Clinical Site, Huntersville, North Carolina
  - Clinical Site, Rock Hill, South Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alizadeh AA, Eisen MB, Davis RE, Ma C, Lossos IS, Rosenwald A, Boldrick JC, Sabet H, Tran T, Yu X, Powell JI, Yang L, Marti GE, Moore T, Hudson J Jr, Lu L, Lewis DB, Tibshirani R, Sherlock G, Chan WC, Greiner TC, Weisenburger DD, Armitage JO, Warnke R, Levy R, Wilson W, Grever MR, Byrd JC, Botstein D, Brown PO, Staudt LM. Distinct types of diffuse large B-cell lymphoma identified by gene expression profiling. Nature. 2000 Feb 3;403(6769):503-11. doi: 10.1038/35000501. PMID 10676951
- [Background] Guinney J, Dienstmann R, Wang X, de Reynies A, Schlicker A, Soneson C, Marisa L, Roepman P, Nyamundanda G, Angelino P, Bot BM, Morris JS, Simon IM, Gerster S, Fessler E, De Sousa E Melo F, Missiaglia E, Ramay H, Barras D, Homicsko K, Maru D, Manyam GC, Broom B, Boige V, Perez-Villamil B, Laderas T, Salazar R, Gray JW, Hanahan D, Tabernero J, Bernards R, Friend SH, Laurent-Puig P, Medema JP, Sadanandam A, Wessels L, Delorenzi M, Kopetz S, Vermeulen L, Tejpar S. The consensus molecular subtypes of colorectal cancer. Nat Med. 2015 Nov;21(11):1350-6. doi: 10.1038/nm.3967. Epub 2015 Oct 12. PMID 26457759
- [Background] Perou CM, Sorlie T, Eisen MB, van de Rijn M, Jeffrey SS, Rees CA, Pollack JR, Ross DT, Johnsen H, Akslen LA, Fluge O, Pergamenschikov A, Williams C, Zhu SX, Lonning PE, Borresen-Dale AL, Brown PO, Botstein D. Molecular portraits of human breast tumours. Nature. 2000 Aug 17;406(6797):747-52. doi: 10.1038/35021093. PMID 10963602
- [Background] Davies H, Bignell GR, Cox C, Stephens P, Edkins S, Clegg S, Teague J, Woffendin H, Garnett MJ, Bottomley W, Davis N, Dicks E, Ewing R, Floyd Y, Gray K, Hall S, Hawes R, Hughes J, Kosmidou V, Menzies A, Mould C, Parker A, Stevens C, Watt S, Hooper S, Wilson R, Jayatilake H, Gusterson BA, Cooper C, Shipley J, Hargrave D, Pritchard-Jones K, Maitland N, Chenevix-Trench G, Riggins GJ, Bigner DD, Palmieri G, Cossu A, Flanagan A, Nicholson A, Ho JW, Leung SY, Yuen ST, Weber BL, Seigler HF, Darrow TL, Paterson H, Marais R, Marshall CJ, Wooster R, Stratton MR, Futreal PA. Mutations of the BRAF gene in human cancer. Nature. 2002 Jun 27;417(6892):949-54. doi: 10.1038/nature00766. Epub 2002 Jun 9. PMID 12068308
- [Background] Schwaederle M, Zhao M, Lee JJ, Lazar V, Leyland-Jones B, Schilsky RL, Mendelsohn J, Kurzrock R. Association of Biomarker-Based Treatment Strategies With Response Rates and Progression-Free Survival in Refractory Malignant Neoplasms: A Meta-analysis. JAMA Oncol. 2016 Nov 1;2(11):1452-1459. doi: 10.1001/jamaoncol.2016.2129. PMID 27273579
- [Background] McShane LM, Cavenagh MM, Lively TG, Eberhard DA, Bigbee WL, Williams PM, Mesirov JP, Polley MY, Kim KY, Tricoli JV, Taylor JM, Shuman DJ, Simon RM, Doroshow JH, Conley BA. Criteria for the use of omics-based predictors in clinical trials. Nature. 2013 Oct 17;502(7471):317-20. doi: 10.1038/nature12564. PMID 24132288
- [Background] McShane LM, Polley MY. Development of omics-based clinical tests for prognosis and therapy selection: the challenge of achieving statistical robustness and clinical utility. Clin Trials. 2013 Oct;10(5):653-65. doi: 10.1177/1740774513499458. Epub 2013 Sep 2. PMID 24000377
- [Background] Lee CH, Yoon HJ. Medical big data: promise and challenges. Kidney Res Clin Pract. 2017 Mar;36(1):3-11. doi: 10.23876/j.krcp.2017.36.1.3. Epub 2017 Mar 31. PMID 28392994
- [Background] Genevieve LD, Martani A, Shaw D, Elger BS, Wangmo T. Structural racism in precision medicine: leaving no one behind. BMC Med Ethics. 2020 Feb 19;21(1):17. doi: 10.1186/s12910-020-0457-8. PMID 32075640
- [Background] Awasthi S, Berglund A, Abraham-Miranda J, Rounbehler RJ, Kensler K, Serna A, Vidal A, You S, Freeman MR, Davicioni E, Liu Y, Karnes RJ, Klein EA, Den RB, Trock BJ, Campbell JD, Einstein DJ, Gupta R, Balk S, Lal P, Park JY, Cleveland JL, Rebbeck TR, Freedland SJ, Yamoah K. Comparative Genomics Reveals Distinct Immune-oncologic Pathways in African American Men with Prostate Cancer. Clin Cancer Res. 2021 Jan 1;27(1):320-329. doi: 10.1158/1078-0432.CCR-20-2925. Epub 2020 Oct 9. PMID 33037017
- [Background] Bentley AR, Callier S, Rotimi CN. Diversity and inclusion in genomic research: why the uneven progress? J Community Genet. 2017 Oct;8(4):255-266. doi: 10.1007/s12687-017-0316-6. Epub 2017 Jul 18. PMID 28770442
- [Background] O'Donnell PH, Dolan ME. Cancer pharmacoethnicity: ethnic differences in susceptibility to the effects of chemotherapy. Clin Cancer Res. 2009 Aug 1;15(15):4806-14. doi: 10.1158/1078-0432.CCR-09-0344. Epub 2009 Jul 21. PMID 19622575
- [Background] Shaw DM, Elger BS, Colledge F. What is a biobank? Differing definitions among biobank stakeholders. Clin Genet. 2014 Mar;85(3):223-7. doi: 10.1111/cge.12268. Epub 2013 Oct 16. PMID 24001330
- [Background] UK Biobank data on 500,000 people paves way to precision medicine. Nature. 2018 Oct;562(7726):163-164. doi: 10.1038/d41586-018-06950-9. No abstract available. PMID 30365879
- [Background] Tutton R. Biobanks and the inclusion of racial/ethnic minorities. Race/ Ethnicity: Multidisciplinary Global Contexts; 2009. p. 75-95.
- See also: National Cancer Institute. Cancer statistics (2018) — https://www.cancer.gov/about-cancer/understanding/statistics
- See also: National Cancer Institute. Cancer types (2018) — https://www.cancer.gov/types
- See also: Jessica Kent. Health Affairs. Accessed December 25, 2020 — https://healthitanalytics.com/news/can-genomic-data-reduce-racial-disparities-in-cancer-outcomes
- See also: Giorgio Sirugo et al, The Missing Diversity in Human Genetic Studies. Cell. Accessed December 25, 2020 — https://doi.org/10.1016/j.cell.2019.02.048